CLINICAL TRIAL: NCT00625690
Title: Development of a Lung Cancer-Screening Program at the University of Nebraska Medical Center: A Feasibility Study
Brief Title: CT Scans in Screening for Lung Cancer in Current and Former Smokers
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0064-05-FB; P30CA036727 (NIH)
Record Dates: First submitted 2008-02-27; First posted 2008-02-28 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of blood sample: At the time of the initial CT scan, every subject will be asked to donate a small blood sample, approximately 10 ml in a yellow EDTA tube (less than 1 tablespoon) from their arm by standard blood drawing techniques, for storage for use in future studies. The blood sample will be number coded, and serum from the blood sample will be stored frozen and held at UNMC for future studies. All studies will be proposed in future IRB submissions.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire administration — Subjects will be asked to complete an additional detailed questionnaire regarding personal information about themselves, their medical history, their diet and lifestyle habits, any past or current environmental exposures and to re-create their family tree for any cancers that have occurred in any of their family members.
Procedure: computed tomography — The baseline and repeat screening CT scans will be performed with a multi-slice helical CT scanner (8 or more rows), at a low-dose setting (120kVp, 40-80mA, slice thickness of 1.25 mm or less). In a single breath-hold, contiguous slices from the thoracic inlet to the adrenal glands will be obtained. Contrast material will not be used. Multi-slice scanners will be used because they provide higher-resolution images. Diagnostic studies, including HRCT will be performed with a multi-slice helical CT at diagnostic settings (120kVp, 140-300mA, slice thickness of 1.25 or less) with the nodule retrospectively reconstructed at a 15cm field of view.
Procedure: evaluation of cancer risk factors — When the CT scan at baseline does not lead to the diagnosis of malignancy, repeat screening will be scheduled 12 months later. If the initial scan led to further evaluation, the repeat scan will be performed 12 months after the most recent scan. The subjects will be allowed to add relevant health information to their record in the web-based database as it develops. Similarly, when in the first repeat screening malignancy is not diagnosed; the second repeat screening will be scheduled 12 months later for a total period of 5 years.
Procedure: study of high risk factors — When the CT scan at baseline does not lead to the diagnosis of malignancy, repeat screening will be scheduled 12 months later. If the initial scan led to further evaluation, the repeat scan will be performed 12 months after the most recent scan. The subjects will be allowed to add relevant health information to their record in the web-based database as it develops. Similarly, when in the first repeat screening malignancy is not diagnosed; the second repeat screening will be scheduled 12 months later for a total period of 5 years.

SUMMARY:
RATIONALE: Screening tests, such as CT scanning, may help doctors find cancer cells early and plan better treatment for lung cancer.

PURPOSE: This clinical trial is studying how well a lung cancer screening program using CT scanning works in current and former smokers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the feasibility of establishing a lung cancer screening program at the University of Nebraska Medical Center using CT scanning in normal study participants with at least a 30 pack-year history of cigarette smoking.
* To determine if it is possible to screen 100 high-risk individuals with high-resolution CT scanning for the presence of suspicious pulmonary nodules.
* To compare an effective and definitive work-up on all study participants with abnormal results within a defined time period from initial screening.

OUTLINE: Study participants complete a detailed questionnaire (paper or electronic version) at baseline to provide personal and family information for inclusion in the registry database. Registry data includes information on participants' medical history, diet, lifestyle habits, and any past or current environmental exposures, as well as family history of cancer within each participant's extended family tree. An instruction manual on completing the questionnaires is provided to all study participants. The System Coordinator of the registry may provide additional information or clarification of the information provided in the questionnaires via a structured telephone interview. Data on study participants and their families is entered into the registry database either manually via the paper-based questionnaires or electronically via interactive Web-based questionnaires completed by participants through the registry website.

Study participants also undergo a low-dose spiral CT scan at baseline. The resulting images are stored electronically and linked to the web-based participant registry. A radiologist then reviews the images, reports on any abnormalities, and renders an interpretation of the scan as being positive or negative for lung nodules. The radiologist's findings are then conveyed to the study participant's primary care physician and the following determinations are made: participants with negative findings (i.e., non-calcified solid nodules < 5 mm or non-solid nodules < 8 mm) are returned home and scheduled for a repeat CT scan in 1 year; participants with abnormalities not related to lung cancer are referred to their primary care physician for further action; and participants with positive findings undergo additional diagnostic work-up and treatment* as described below.

* Non-calcified solid nodules ≥ 5 and ≤ 15 mm: Study participants undergo a course of antibiotics followed by a high-resolution CT scan at 3 months. If the CT findings are stable, then participants return for a repeat CT scan in 1 year. If the nodules are growing, participants undergo additional diagnostic work-up, which may include biopsy of the positive nodule by their treating clinician.
* Non-solid nodule ≥ 8 mm: Study participants undergo treatment with an antibiotic, CT follow-up, and additional diagnostic work-up, if appropriate, as described previously.
* Non-calcified solid nodules > 15 mm: Study participants undergo work-up for a positive nodule, as above.

NOTE: *Study participants who demonstrate radiographic abnormalities that are suspected to be of an inflammatory nature are given a 10-day course of a broad spectrum respiratory antibiotic, preferably a fluoroquinolone, by the participating physician who enrolled that participant into the study.

Study participants with negative CT findings undergo CT screening once yearly for up to five years, in the absence of a diagnosed malignancy. Diagnostic work-up for repeat CT scans is as follows:

* Any new lesion: Study participants undergo a work-up as previously described for non-calcified solid or non-solid nodules.
* Any non-calcified nodule that was present earlier and grew in size:

  * Growth < 3 mm: Study participants undergo a repeat CT scan in 6 months. If there is further growth, participants are worked-up for a positive nodule, or, if the scan is stable, participants undergo a repeat scan 1 year after the most recent scan.
  * Growth between 3 mm and 5 mm: Study participants undergo a high-resolution CT scan in 3 months and further diagnostic work-up for a positive nodule, as described previously, if there is growth. If there is complete resolution of the nodule, participants undergo repeat screening CT scan in 1 year after the most recent scan. If there is partial resolution of the nodule, another high-resolution CT scan is performed 3 months later. Participants with a stable nodule undergo repeat screening CT scan 1 year after the most recent scan.
  * Growth ≥ 5 mm: Study participants receive a course of an antibiotic and undergo high-resolution CT scanning after 1 month. The following assessments are also performed: work-up for a positive nodule, if there is further growth; repeat screening CT scan in 1 year after the most recent scan, if there is complete resolution of the nodule; high-resolution CT scan in 3 months, if there is partial resolution of the nodule; and repeat screening CT scan 1 year after the most recent scan, if the nodule is stable.

All study participants undergo blood sample collection at baseline for use in future studies. Additional blood samples are obtained from study participants with positive CT scans for future research on smoking-related diseases. Tissue samples obtained from diagnostic biopsy or surgical specimens are also stored for future research.

Once a malignancy is diagnosed and a definitive intervention is performed, study participants are followed periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Current and former smokers with at least a 30 pack-year history of smoking
* Body weight less than 140 kg (308 pounds)
* Able to lie flat
* Able to comply with long-term follow-up
* Functional capacity and willingness to undergo diagnostic work-up of suspicious nodules and curative therapy if lung cancer is detected
* Nursing mothers allowed
* Able to come to clinic for screening

Exclusion Criteria:

* No cognitive impairment that would preclude providing informed consent
* No other concurrent or prior malignancy within the past five years except superficial basal cell carcinoma or nonmelanoma skin cancer
* No condition that would preclude screening, diagnosis, or surgical treatment
* Not pregnant/negative pregnancy test

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Normal subjects with at least a 30 pack-year history of cigarette smoking.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-05-19 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of establishing a lung cancer screening program at the University of Nebraska Medical Center | Upon the approximately 5-year establishment of normative parameters in regard to screening efficiency.
  Frequency of suspicious nodules on baseline CT; Frequency of invasive procedures for diagnosis; Frequency of surgical evaluation; Complication rates with diagnostic work up as well as surgical management.
Feasibility of screening 100 high-risk individuals with high-resolution CT scanning for the presence of suspicious pulmonary nodules | Upon the approximately 5-year establishment of normative parameters in regard to screening efficiency.
  Enrollment of 100 subjects; Baseline and yearly CT evaluations for 4 more years.
Comparison of work-up on all study participants with abnormal results within a defined time period from initial screening | Upon the approximately 5-year establishment of normative parameters in regard to screening efficiency.
  Participants with abnormalities not related to lung cancer are referred to their primary care physician for further action; and participants with positive findings undergo additional diagnostic work-up and treatment. NOTE: Study participants who demonstrate radiographic abnormalities that are suspected to be of an inflammatory nature are given a 10-day course of a broad spectrum respiratory antibiotic, preferably a fluoroquinolone, by the participating physician who enrolled that participant into the study.
Frequency of suspicious nodules at baseline | Upon the approximately 5-year establishment of normative parameters.
  Study participants undergo a low-dose spiral CT scan at baseline. A radiologist then reviews the images, reports on any abnormalities, and renders an interpretation of the scan as being positive or negative for lung nodules. The radiologist's findings are then conveyed to the study participant's primary care physician.
Frequency of invasive procedures for diagnosis | Upon the approximately 5-year establishment of normative parameters.
  Non-calcified solid nodules ≥ 5 and ≤ 15 mm: If the nodules are growing, participants undergo additional diagnostic work-up, which may include biopsy of the positive nodule by their treating clinician.
  Non-solid nodule ≥ 8 mm: Additional diagnostic work-up, if appropriate, as described previously.
  Non-calcified solid nodules > 15 mm: Work-up for a positive nodule, as above.
Frequency of surgical evaluation | Upon the approximately 5-year establishment of normative parameters
  Non-calcified solid nodules ≥ 5 and ≤ 15 mm: If the nodules are growing, participants undergo additional diagnostic work-up, which may include biopsy of the positive nodule by their treating clinician.
  Non-solid nodule ≥ 8 mm: Additional diagnostic work-up, if appropriate, as described previously.
  Non-calcified solid nodules > 15 mm: Work-up for a positive nodule, as above.
Complication rates with diagnostic work-up | Upon the approximately 5-year establishment of normative parameters.
  All study participants undergo blood sample collection at baseline for use in future studies. Additional blood samples are obtained from study participants with positive CT scans for future research on smoking-related diseases. Tissue samples obtained from diagnostic biopsy or surgical specimens are also stored for future research.
Surgical management | Upon the approximately 5-year establishment of normative parameters.
  If malignancy is diagnosed, that patient after definitive intervention will be followed for progression-free survival and cancer-related mortality. In case the subject develops any malignancy, the subject will be taken off study but the course of the malignancy, including survival will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Apar K Ganti, MD, Principal Investigator — University of Nebraska
Locations (1):
- Eppley Cancer Center, University of Nebraska Medical Center, Omaha, Nebraska, United States